CLINICAL TRIAL: NCT03209791
Title: Mechanisms of Skeletal Muscle Proteolysis With Ethanol Consumption: an Integrated Molecular Metabolic Approach
Brief Title: Ethanol Induces Skeletal Muscle Autophagy
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Other Study IDs: 14-1287
Record Dates: First submitted 2017-04-14; First posted 2017-07-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Alcoholic Steatosis: This group will have 10 patients with alcoholic steatosis which is milder disease and muscle biopsies will be performed
  Interventions: Other: Biopsies
- Cirrhosis: This group will consist of 10 patients with cirrhosis. We anticipate a 50% difference in these patients and the controls in the autophagy readouts and muscle biopsies will be performed
  Interventions: Other: Biopsies
- Steatohepatitis: This group will have 10 patients with alcoholic steatohepatitis that have more severe necroinflammation in the liver but for a shorter duration of illness and muscle biopsies will be performed
  Interventions: Other: Biopsies
- controls: This group will consist of 10 patients who are healthy and have no liver disease diagnosis and muscle biopsies will be performed
  Interventions: Other: Biopsies

INTERVENTIONS:
Other: Biopsies — Biopsy will be done on the Vastus Lateralis muscle in all groups

SUMMARY:
In this study we plan to demonstrate that ethanol induces skeletal muscle autophagy to degrade MAA adducts.

DETAILED DESCRIPTION:
Hypothesis: Ethanol mediated modification of skeletal muscle proteins to form MAA adducts that in turn induce skeletal muscle autophagy.

Patients with alcoholic steatosis, hepatitis and cirrhosis (n=10 each) will be recruited from the liver transplant nutrition clinic or the hepatology inpatient service and their body composition quantified using anthropometry, bioelectrical impedance analysis, CT image analysis and DEXA if available.

Control Subjects. Controls will be recruited by advertisement. All control subjects will have a normal clinical history, physical examination, and screening chemistries. They will not have any significant medical conditions requiring the use of medications. Their nutritional status within 20% of normal as defined by ideal body weight.

ELIGIBILITY:
Inclusion Criteria:

Alcoholic liver disease:

* clinical, biochemical, imaging criteria and liver biopsy where available
* Age 18 - 65 years old

Controls:

* Serum liver transaminases (i.e. ALT and AST) 40 IU/L
* Normal liver ultrasound
* Age 18 - 65 years old

Exclusion Criteria:

For both groups - alcoholic liver disease and controls:

* Poorly controlled diabetes mellitus (HbA1C>9.5 g/dl)
* Untreated Hyper- / hypo- thyroidism
* Patients on dialysis, renal disease with serum creatinine 1.5 mg/dL
* Active intravenous drug use
* History of bowel surgery or gastric bypass surgery
* Medications known to alter muscle protein metabolism (i.e. corticosteroids, tamoxifen, high-dose estrogen, testosterone or anabolic steroids)
* Metastatic disease, Advanced cardiac or pulmonary disease
* Pregnancy
* Coagulopathy- INR >1.4 and platelet count <80,000/ml.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Histologically characterized patients with alcoholic steatosis, hepatitis and cirrhosis (n=10 each) will be recruited from the liver transplant nutrition clinic or the hepatology inpatient service and their body composition quantified using protocols already established by the PI.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-05-18 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Autophagy | 4 hours
  We will measure Malonyldialdehyde Acetaldehyde protein adducts to see skeletal muscle proteolysis during a one time muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Dasarathy, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No